CLINICAL TRIAL: NCT00552539
Title: Video Tool to Promote Syphilis Knowledge and Testing in the Emergency Department
Brief Title: Syphilis Video Tool to Promote Knowledge and Testing in the ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacobi Medical Center (Other)
Collaborators: Public Health Solutions (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 06431
Record Dates: First submitted 2007-10-31; First posted 2007-11-02 (Estimated); Last update posted 2007-11-02 (Estimated); Status verified 2007-10

CONDITIONS: Syphilis
Keywords: syphilis; educational video; knowledge; black; Hispanic
MeSH Terms: conditions — Syphilis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): pre test survey, educational video, post test survey
  Interventions: Other: 'educational video'
- 2 (No Intervention): no intervention
- 3 (Experimental): educational video and post test survey
  Interventions: Other: 'educational video'
- 4 (No Intervention): post test survey

INTERVENTIONS:
Other: 'educational video' — 'educational video'
  Arms: 1; 3

SUMMARY:
The objective of this study is to determine whether the "Syphilis and Men" educational video can be a useful tool to increase syphilis knowledge and testing among English and Spanish-speaking urgent care and emergency department patients, regardless of various self-reported characteristics that increase their risk for syphilis infection.

DETAILED DESCRIPTION:
A randomized four-group intervention-control Solomon design was implemented with Group 1 participants receiving a pre-test survey, the educational video intervention, and a post-test survey; Group 2 the pre-test and post-test surveys; Group 3 the video intervention and a post-test survey; and Group 4 the post-test survey. This design was selected to assess the effect of the video in increasing syphilis knowledge while controlling for the influence of the pre-test instrument in potentially sensitizing participants to key facts. A computer-generated randomization list was created and used to assign patients to groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-55 years of age were eligible only if they spoke English or Spanish.

Exclusion Criteria:

* Patients were excluded if clinically unstable, unarousable, hearing impaired or visually impaired despite corrected lens.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2006-06; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
The primary outcome was the score on a 10-question measure designed to assess knowledge attained from the educational video. | 20 minutes

SECONDARY OUTCOMES:
A secondary outcome was the decision to be tested for syphilis. | 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Yvette Calderon, MD, MS, Principal Investigator — Jacobi Medical Center; John P Sanchez, MD, MPH, Principal Investigator — Jacobi Medical Center
Locations (1):
- Jacobi Medical Center, The Bronx, New York, United States